CLINICAL TRIAL: NCT04975503
Title: Classical Risk Factors in Young Middle Eastern Women With Atherosclerotic Cardiovascular Disease
Brief Title: Risk Factors in Young Middle Eastern Women With Cardiovascular Disease
Status: Completed | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Principal Investigator, Ayman J Hammoudeh, MD, FACC, Interventional Cardiologist, Department of cardiology, Istishari Hospital, Amman, Jordan, Jordan Collaborating Cardiology Group
Other Study IDs: IH/JCCG1-RFYW
Record Dates: First submitted 2021-07-14; First posted 2021-07-23 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Cardiovascular Diseases; Risk Factors
Keywords: Atherosclerotic cardiovascular disease; Risk factors
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young Women: Young women, aged 18 to 50 years, with documented atherosclerotic cardiovascular disease
  Interventions: Other: Observing cardiovascular risk factors
- Older Women: Older women, aged >50 years, with documented atherosclerotic cardiovascular disease
  Interventions: Other: Observing cardiovascular risk factors

INTERVENTIONS:
Other: Observing cardiovascular risk factors — Documenting the presence or absence of CVD risk factors in each participant.

SUMMARY:
Cardiovascular disease continues to be the leading cause of death among women in the Middle East, including Jordan. Sex-specific data focused on cardiovascular disease have been increasing steadily, yet is not the subgroup of young women. This study focuses on classical and novel risk factors of cardiovascular disease in young women compared with older women.

DETAILED DESCRIPTION:
This is the introduction of a new study at Istishari entitled: "The Classical Risk Factors in Young Middle Eastern Women with Atherosclerotic Cardiovascular Disease" This is an investigator-initiated, cross-sectional, non-interventional, observational study.

Medical research in Jordan is a basic responsibility of all medical sectors in the country. Despite the drastic growth and advances of medical services, the volume of the local medical research is, at best estimate, scarce. The emerging role of private medical groups, private hospitals, and residency programs in cooperation with other medical sectors and medical schools, in conducting, presenting, and publishing such studies should be encouraged and supported. A major indicator of judging the credibility and quality of any medical research project is to look at the conferences the research was presented at and the journals it was published in.

This is the 10th major project of the Jordan Collaborating Cardiology Group (JCC) and the first in cooperation with the Istishari Hospital Internal Medicine Residency Program (see Appendix 1. Timeline of JCC Group studies) The first project was JoHARTS that evaluated coronary risk factors and dyslipidemia in 5000 individuals with ACS, stable CAD, and non CAD patients. The 2nd project was CAPRIS evaluated the prognostic implications of hs-CRP in ACS from admission to 1 year. The 3rd project was MINTOR that evaluated onset, triggers, reperfusion strategies, and hospital mortality in more than 950 Jordanians with acute ST-elevation MI. The 4th project was GLORY study that evaluated the prevalence of glucometabolic states among ACS patients, prognosis up to 1 year, and TIMI risk score . The 5th was JoPCR1 that evaluated outcome post PCI in 2426 ACS and non ACS patients in 12 tertiary care centers for the incidence of death, stent thrombosis, revascularization, bleeding, impact of gender, DM, renal dysfunction, and age on outcome, GRACE, and CRUSADE risk scores. The 6th is the colchicine study of AF prevention in open heart surgery, one is completed with 1 mg dose and one is ongoing with reduced dose. The 7th and 8th projects are ongoing and study statin eligibility in patients admitted with MI (Statin EPIC) and decade or more survivors after coronary revascularization. The 8th was the Jordanian AF study which evaluated patients with AF in ambulatory and out-patient settings. The 9th was the JoCORE study that evaluated acute CV events due to the stresses of the covid-19 pandemic.

One population subgroup is under studied in the world literature as well as the local literature. The young women who have documented CVD. This group represents only a small proportion of the CVD population in all countries.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 y or more.
* Documented CVD (CAD stable or ACS, PCI, CABG, CVA/TIA, carotid disease, PAD).

Exclusion Criteria:

* Women younger than 18 years of age.
* No documented CVD.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Study Population: The prevalence of the 4 classical risk factors (HTN, DM, smoking, and dyslipidemia) will be studied in young women (younger than 50 years of age, and older than 18 y of age) who have documented CVD in ambulatory and in-patient settings.
  This data will be compared with those from women older than 50 y of age with CVD.
Sampling Method: Non-Probability Sample
Enrollment: 627 (Actual)
Dates: Start 2021-08-22 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of classical CVD risk factors | August 2021 to September 2020.
  To study the prevalence of the 4 classical risk factors (HTN, DM, smoking, and dyslipidemia) in young women (younger than 50 years of age) who have documented CVD in ambulatory and in-patient settings and compare the data with women older than 50 y of age with CVD.

SECONDARY OUTCOMES:
Prevalence of novel/emerging CVD risk factors | August 2021 to September 2022.
  To study emerging non traditional risk factors, and demographic baseline features of these patients including family history, BMI, PCOS, hormone medications, sport activities.. etc.

CONTACTS AND LOCATIONS:
Overall Officials: Reham Nasseddin, MD, Study Director — Jordan Collaborating Cardiology Group; Laith N Habahbeh, MD, Study Director — Jordan Collaborating Cardiology Group
Locations (1):
- Istishari Hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: No
The individual participant data will be retained with the PI and not shared. Clinical forms with participant initials, rather than full names, will be shared for analysis.

REFERENCES:
- [Derived] Hammoudeh AJ, Jallad M, Khader Y, Badaineh Y, Tabbalat RA, Zammar H, Al-Makhamreh H, Basha A, AlAtteili L, Abuhalimeh R, Fkheideh T, Ababneh A, Ababneh L, Mahmoud SA, Alhaddad IA. Atherosclerotic Cardiovascular Disease Novel and Traditional Risk Factors in Middle Eastern Young Women. The ANCORS-YW Study. Glob Heart. 2024 Jul 15;19(1):59. doi: 10.5334/gh.1341. eCollection 2024. PMID 39035774